CLINICAL TRIAL: NCT00654420
Title: An Open Label, Randomized Phase I/IIa Trial Evaluating MK-0646 in Combination With Erlotinib (TARCEVA™) for Patients With Recurrent Non-Small Cell Lung Cancer
Brief Title: A Study Evaluating Dalotuzumab (MK-0646) in Combination With Erlotinib for Participants With Non-Small Cell Lung Cancer (MK-0646-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0646-007; 2007_605 (Other: Merck Registration Number); 2007-005941-39 (EudraCT Number)
Record Dates: First submitted 2008-03-26; First posted 2008-04-08 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma, Non-small-cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dalotuzumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ph I: Dalotuzumab 5 mg/kg + Erlotinib (Experimental): During the Phase I part of the study, participants receive dalotuzumab intravenously (IV) at 5 mg/kg weekly plus open-label erlotinib at 150 mg daily for 4 weeks. After 4 weeks of therapy, participants in Phase I who do not have disease progression and are satisfactorily tolerating study drug can continue to receive study drug.
  Interventions: Drug: Dalotuzumab
- Ph I: Dalotuzumab 10 mg/kg + Erlotinib (Experimental): During the Phase I part of the study, participants receive dalotuzumab intravenously (IV) at 10 mg/kg weekly plus open-label erlotinib at 150 mg daily for 4 weeks. After 4 weeks of therapy, participants in Phase I who do not have disease progression and are satisfactorily tolerating study drug can continue to receive study drug.
  Interventions: Drug: Dalotuzumab
- Ph II: Dalotuzumab 10 mg/kg + Erlotinib (Experimental): During the Phase II part of the study, participants are randomized to receive dalotuzumab intravenously (IV) at 10 mg/kg weekly plus open-label erlotinib at 150 mg daily until disease progression or occurrence of unacceptable toxic effects.
  Interventions: Drug: Dalotuzumab
- Ph II: Erlotinib (Active Comparator): During the Phase II part of the study, participants are randomized to receive open-label erlotinib at 150 mg daily until disease progression or occurrence of unacceptable toxic effects.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Dalotuzumab — Dalotuzumab 20 mg/mL in sterile solution. Intravenous (IV) infusion over 60 minutes at 5 mg/kg, administered weekly at dosage according to treatment group.
  Other Names: MK-0646
  Arms: Ph I: Dalotuzumab 10 mg/kg + Erlotinib; Ph I: Dalotuzumab 5 mg/kg + Erlotinib; Ph II: Dalotuzumab 10 mg/kg + Erlotinib
Drug: Erlotinib — Open-label erlotinib administrated orally (tablets) by mouth (PO) at 150 mg daily.
  Other Names: Tarceva; Erlotinib hydrochloride
  Arms: Ph II: Erlotinib

SUMMARY:
This is a Phase I/IIa study to evaluate safety and efficacy of dalotuzumab (MK-0646) in combination with erlotinib in participants with recurrent Non-Small Cell Lung Cancer (NSCLC). The Phase I part of this study will determine the highest tolerated dose of dalotuzumab to be given in combination with erlotinib. The primary hypothesis for the Phase I part of the study is that administration of erlotinib in combination with dalotuzumab in participants with recurrent NSCLC is generally well-tolerated as evidenced by accumulated safety data from this trial. The Phase II part of this study will investigate how well dalotuzumab works in conjunction with erlotinib at treating recurrent NSCLC. The primary hypothesis for the Phase II part of this study is that administration of erlotinib in combination with dalotuzumab in participants with recurrent NSCLC results in improvement in Progression Free Survival (PFS) compared to participants treated with erlotinib alone. PFS is defined as the time from randomization until either the emergence of radiographic evidence of disease progression (as documented by an independent core laboratory) or death due to any cause, whichever occurs first.

DETAILED DESCRIPTION:
Dalotuzumab is a humanized monoclonal antibody (mAb) that targets the Insulin-like Growth Factor Receptor (IGF-1R). Dalotuzumab may act through:

* Inhibition of IGF-1-mediated cell signaling to cause reductions in tumor growth and spread
* Antibody dependent cell-mediated cytotoxicity

In preclinical studies, dalotuzumab improved the activity of an anti-Epidermal Growth Factor Receptor (EGFR) mAb and the activity of Erlotinib, a small molecule inhibitor of EGFR

Trial Duration of Treatment: Participants will continue on the study for as long as their disease is not progressing and they do not have unmanageable side effects from the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant has locally advanced or metastatic stage IIIB/IV NSCLC that has relapsed after hemotherapy/chemoratiotherapy
* Participant has had at least one chemotherapy regimen for recurrent or metastatic disease
* Participant is 18 years of age or older
* Participant has a performance status of 0-2 on Eastern Cooperative Group (ECOG) scale
* Women of childbearing potential have a negative pregnancy test

Exclusion Criteria:

* Participant has had chemotherapy within 2 weeks or biological therapy (e.g. bevacizumab) within 4 weeks
* Participant has not recovered from adverse events from previous therapy within 4 weeks
* Participant has received EGFR-Tyrosine Kinase Inhibitor (TKI) inhibitor/anti-EGFR mAb therapy
* Participant has received IGF1R-TKI inhibitor/anti-IGF1R mAB therapy
* Participant has had more than 2 systemic chemotherapies for metastatic disease
* Participant has not completed radiotherapy with complete resolution of toxicities at least 2 weeks before starting in the study
* Participant is taking part in another clinical study
* Participant has a primary central nervous system tumor
* Participant abuses drugs or alcohol
* Participant is pregnant or breastfeeding
* Participant is Human Immunodeficiency Virus (HIV) positive
* Participant has a history of hepatitis B or C
* Participant is using growth hormone or growth hormone inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-03-19 (Actual); Primary Completion 2009-11-25 (Actual); Study Completion 2012-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Moran T, Felip E, Keedy V, Borghaei H, Shepherd FA, Insa A, Brown H, Fitzgerald T, Sathyanarayanan S, Reilly JF, Mauro D, Hsu K, Yan L, Johnson DH. Activity of dalotuzumab, a selective anti-IGF1R antibody, in combination with erlotinib in unselected patients with Non-small-cell lung cancer: a phase I/II randomized trial. Exp Hematol Oncol. 2014 Nov 7;3(1):26. doi: 10.1186/2162-3619-3-26. eCollection 2014. PMID 25414803
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/study.html?id=0646-007&kw=0646-007&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 participants were enrolled in Phase I part (dose escalation) and 75 participants were enrolled in Phase II part of study (95 total enrolled).
Groups:
- Ph I: Dalotuzumab 5 mg/kg + Erlotinib: During the Phase I part of the study, participants received dalotuzumab intravenously (IV) at 5 mg/kg weekly plus open-label erlotinib at 150 mg daily for 4 weeks. After 4 weeks of therapy, participants in Phase I who did not have disease progression and were satisfactorily tolerating study drug could continue to receive study drug.
- Ph I: Dalotuzumab 10 mg/kg + Erlotinib: During the Phase I part of the study, participants received dalotuzumab IV at 10 mg/kg weekly plus open-label erlotinib at 150 mg daily for 4 weeks. After 4 weeks of therapy, participants in Phase I who did not have disease progression and were satisfactorily tolerating study drug could continue to receive study drug.
- Ph II: Dalotuzumab 10 mg/kg + Erlotinib: During the Phase II part of the study, participants were randomized to receive dalotuzumab IV at 10 mg/kg weekly plus open-label erlotinib at 150 mg daily until disease progression or occurrence of unacceptable toxic effects.
- Ph II: Erlotinib: During the Phase II part of the study, participants were randomized to receive open-label erlotinib at 150 mg daily until disease progression or occurrence of unacceptable toxic effects.
Period: Phase I (Dose Escalation)
Arm/Group | Ph I: Dalotuzumab 5 mg/kg + Erlotinib | Ph I: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Erlotinib
Started | 4 | 16 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 16 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 4 | 15 | 0 | 0
Period: Phase II
Arm/Group | Ph I: Dalotuzumab 5 mg/kg + Erlotinib | Ph I: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Erlotinib
Started | 0 | 0 | 37 (New participants were enrolled in the Phase II part of the study that did not participate in Phase 1) | 38 (New participants were enrolled in the Phase II part of the study that did not participate in Phase 1)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 37 | 38
Not completed — Adverse Event | 0 | 0 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 4
Not completed — Progressive Disease | 0 | 0 | 29 | 29
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 1
Not completed — Missing Disposition Record | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ph I: Dalotuzumab 5 mg/kg + Erlotinib: During the Phase I part of the study, participants received dalotuzumab IV at 5 mg/kg weekly plus open-label erlotinib at 150 mg daily for 4 weeks. After 4 weeks of therapy, participants in Phase I who did not have disease progression and were satisfactorily tolerating study drug could continue to receive study drug.
- Total: Total of all reporting groups
Arm/Group | Ph I: Dalotuzumab 5 mg/kg + Erlotinib | Ph I: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Erlotinib | Total
Number analyzed (Participants) | 4 | 16 | 37 | 38 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (3.86) | 61.9 (7.68) | 61.9 (7.83) | 58.5 (10.35) | 60.2 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 10 | 10 | 22
  Male | 4 | 14 | 27 | 28 | 73

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants Experiencing at Least One Dose-Limiting Toxicity (DLT) Adverse Event (AE) During the First Four Weeks of Dalotuzumab Plus Erlotinib Treatment
Description: A DLT was an AE related (definitely, probably, or possibly) to study therapy and occurring within first 4 weeks of therapy.
  Hematologic DLTs included Grade (Gr)4 neutropenia lasting for ≥7 days, Gr 3/Gr 4 neutropenia with fever >38.5 °C and/or infection requiring antibiotic or anti-fungal treatment, and Gr 4 thrombocytopenia (25.0 x 10^9/L).
  Non-hematologic DLT defined as any ≥Gr 3 nonhematologic toxicity, except Gr 3 reversible rash; Gr 3 nausea, vomiting, diarrhea, dehydration, or hyperglycemia occurring in setting of inadequate compliance with supportive care; alopecia; anorexia; asthenia; inadequately-treated hypersensitivity reactions; Gr 3 elevated transaminases (≤1 week duration); or infusion reactions to dalotuzumab.
  Any drug-related AEs that led to dose modification of dalotuzumab/erlotinib or any unresolved drug-related toxicity that caused a ≥3 week delay of next scheduled dose of study drug, regardless of Common Terminology Criteria grade, were DLTs.
Time Frame: Up to 4 weeks after initiation of treatment
Population: Participants in the Phase I part of the study who received at least one dose of dalotuzumab in combination with erlotinib during the first 4 weeks of treatment and were evaluable for DLT assessment. Participants in the Phase II part of the study were not evaluated for DLTs.
Measure: Number; unit: participants
Arm/Group | Ph I: Dalotuzumab 5 mg/kg + Erlotinib | Ph I: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Erlotinib
Number analyzed (Participants) | 4 | 13 | 0 | 0
participants | 0 | 1 |  |

2. Primary Outcome: Phase II: Median Progression Free Survival (PFS) in Participants Receiving Dalotuzumab Plus Erlotinib Treatment
Description: PFS was defined as the time from randomization until either the emergence of radiographic evidence of disease progression or death due to any cause, whichever occurs first. Disease progression was classified as a radiographic assessment of progressive disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) using computed tomography (CT) or magnetic resonance imaging (MRI). As pre-specified by the protocol, final analysis of PFS was to take place after approximately 49 PFS events or deaths had occurred in the Phase II part of the trial. A non-parametric Kaplan-Meier method was used to estimate the median PFS time for each treatment group. Participants who discontinued from the study for reasons other than progression of disease were treated as right-censored observations at the time of the last response evaluation. Participants who withdrew from the study due to PD were considered to have a disease progression between the last visit and the time of withdrawal.
Time Frame: Duration of time required to collect approximately 49 deaths or PFS events (assessed up to ~20 months total on this study from randomization to cut-off date)
Population: All randomized participants in Phase II who received ≥1 dose of study treatment, had a baseline radiological (CT or MRI) disease assessment, and had ≥1 post-baseline radiological (CT or MRI) disease assessment subsequent to ≥1 dose of study treatment for reason other than discontinuation for AE. Phase I participants were not assessed for PFS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ph I: Dalotuzumab 5 mg/kg + Erlotinib | Ph I: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Erlotinib
Number analyzed (Participants) | 0 | 0 | 36 | 36
months |  |  | 2.5 [1.4 to 5.3] | 1.6 [1.3 to 2.7]
Statistical Analysis 1: Comparison: Ph II: Dalotuzumab 10 mg/kg + Erlotinib vs Ph II: Erlotinib; Finkelstein proportional hazards model for interval-censored data was used to assess treatment effect on PFS in Phase II. The hazard ratio with 95% confidence interval for the Dalotuzumab (10 mg/kg) + Erlotinib treatment arm compared to the Erlotinib treatment arm was reported; Test type: Superiority or Other; p = 0.268, Finkelstein Proportional Hazards Model; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.47 to 1.57]

3. Secondary Outcome: Phase II: Median Overall Survival (OS) in Participants Receiving Dalotuzumab Plus Erlotinib Treatment
Description: OS was defined as the time from randomization to death in months due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. The nonparametric Kaplan-Meier method was used to estimate the survival time distribution and the median survival of each treatment group.
Time Frame: as for outcome 2
Population: Intent to Treat (IIT) Population; all randomized participants in Phase II included regardless of compliance to planned treatment. Phase I participants were not assessed for OS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ph I: Dalotuzumab 5 mg/kg + Erlotinib | Ph I: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Erlotinib
Number analyzed (Participants) | 0 | 0 | 37 | 38
months |  |  | 6.9 [5.2 to 14.7] | 14.5 [8.2 to NA] — A statistical estimate of the upper bound is not available based on the model used for the data analysis.
Statistical Analysis 1: Comparison: Ph II: Dalotuzumab 10 mg/kg + Erlotinib vs Ph II: Erlotinib; The treatment difference in survival between treatment groups was assessed by Cox regression. The estimated hazard ratio for treatment of the Dalotuzumab (10 mg/kg) + Erlotinib treatment arm compared to the Erlotinib treatment arm was reported from the Cox model; Test type: Superiority or Other; p = 0.879, Regression, Cox; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.78 to 2.64]

4. Secondary Outcome: Phase II: Percentage of Participants With Complete Response (CR) or Partial Response (PR) After Dalotuzumab Plus Erlotinib Treatment (Objective Response Rate [ORR])
Description: ORR was defined as the percentage of participants in the Phase II analysis population having complete response (CR) or partial response (PR) during the course of the study.
  RECIST criteria were used to quantify response rate. For evaluation of target lesions, CR was defined as disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of the LD. For evaluation of non-target lesions, CR was defined as disappearance of all non-target lesions and normalization of tumor marker level.
  Confirmation of response required a second assessment performed 4 weeks or more after the initial assessment. If the confirmation assessment contradicted the initial assessment, it was considered that a response had not been observed. If the confirmation assessment of a participant was not available, that participant was not considered as a responder in the response rate analyses.
Time Frame: as for outcome 2
Population: All randomized participants in Phase II who received ≥1 dose of study treatment, had a baseline radiological (CT or MRI) disease assessment, and had ≥1 post-baseline radiological (CT or MRI) disease assessment subsequent to ≥1 dose of study treatment for reason other than discontinuation for AE. Phase I participants were not assessed for ORR.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ph I: Dalotuzumab 5 mg/kg + Erlotinib | Ph I: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Erlotinib
Number analyzed (Participants) | 0 | 0 | 36 | 36
percentage of participants |  |  | 2.8 [0.1 to 14.5] | 5.6 [0.7 to 18.7]
Statistical Analysis 1: Comparison: Ph II: Dalotuzumab 10 mg/kg + Erlotinib vs Ph II: Erlotinib; Miettinen and Nurminen's method for stratified data was used for comparison of percentage of participants with objective response (ORR) between the two treatment groups. Response rate calculation was based on full follow-up; Test type: Superiority or Other; p = 0.721, Miettinen & Nurminen Method; Difference in Percentage = -2.8, 95% CI 2-sided [-15.9 to 9.4]

ADVERSE EVENTS:
Time Frame: Up to 47 months
Description: All Participants as Treated (APaT) population; all allocated participants who received at least one dose of study treatment.
Arm/Group | Ph I: Dalotuzumab 5 mg/kg + Erlotinib | Ph I: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Dalotuzumab 10 mg/kg + Erlotinib | Ph II: Erlotinib
Serious Adverse Events (participants affected / at risk) | 3/4 | 4/16 | 19/37 | 22/38
Other Adverse Events (participants affected / at risk) | 4/4 | 16/16 | 37/37 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph I: Dalotuzumab 5 mg/kg + Erlotinib (N=4) | Ph I: Dalotuzumab 10 mg/kg + Erlotinib (N=16) | Ph II: Dalotuzumab 10 mg/kg + Erlotinib (N=37) | Ph II: Erlotinib (N=38)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 4 (5)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 8 (8) | 5 (6)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph I: Dalotuzumab 5 mg/kg + Erlotinib (N=4) | Ph I: Dalotuzumab 10 mg/kg + Erlotinib (N=16) | Ph II: Dalotuzumab 10 mg/kg + Erlotinib (N=37) | Ph II: Erlotinib (N=38)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 6 (6) | 2 (13)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Trichomegaly (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (9) | 6 (11)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (3) | 4 (6) | 4 (6)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 12 (16) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 11 (49) | 30 (48) | 27 (75)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (3) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 17 (27) | 17 (23)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 5 (7) | 4 (4) | 3 (3)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (7) | 7 (9) | 10 (16)
Asthenia (General disorders) | 1 (1) | 10 (16) | 13 (20) | 13 (26)
Chest pain (General disorders) | 1 (1) | 4 (4) | 2 (2) | 8 (9)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (3) | 11 (15) | 13 (16)
Mucosal inflammation (General disorders) | 3 (4) | 2 (3) | 5 (6) | 3 (3)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (6)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 5 (9) | 5 (9) | 6 (7)
Visceral pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (11) | 1 (1)
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecthyma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 1 (1) | 6 (10) | 8 (10)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 4 (7) | 4 (4)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Blood amylase increased (Investigations) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 3 (8)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 5 (6) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 7 (11) | 22 (26) | 21 (26)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (21) | 6 (8) | 5 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 5 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (5) | 5 (6)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 7 (9) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (5)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 5 (7) | 3 (5)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 3 (3) | 4 (4) | 5 (6)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) | 4 (4)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (5) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 7 (8) | 7 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (8) | 5 (5) | 12 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 4 (5) | 4 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3) | 4 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (4) | 1 (1) | 2 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 3 (3) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (12) | 6 (12) | 3 (4) | 8 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 9 (9) | 7 (10)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5) | 2 (2) | 4 (6)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6) | 7 (10) | 11 (11)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 8 (13) | 28 (45) | 22 (39)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6) | 2 (2) | 7 (8)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.